CLINICAL TRIAL: NCT02750254
Title: A Phase I/II Study of Azacitidine in Haploidentical Donor Hematopoietic Cell Transplantation
Brief Title: Azacitidine in Haploidentical Donor Hematopoietic Cell Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity. Only enrolled patients in phase I portion of trial.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201604081
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; fludarabine phosphate; Busulfan; Cyclophosphamide; Whole-Body Irradiation; Melphalan; Granulocyte Colony-Stimulating Factor; plerixafor; Filgrastim; Stem Cell Transplantation; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Azacitidine (Experimental): * Treating physician must choose from one of these conditioning regimens (will be given per standard of care)
    * fludarabine and fractionated total body irradiation (Flu/FrTBI)
    * fludarabine and busulfan (Flu/Bu4)
    * fludarabine, cyclophosphamide, and single dose total body irradiation (Flu/Cy/sdTBI)
    * fludarabine and melphalan (Flu/Mel)
    * reduced-intensity fludarabine and busulfan (Flu/Bu2)
  * G-CSF from Day -5 through Day -1 per standard of care
  * On Day 0, the allograft will be infused per standard of care.
  * Azacitidine will be administered on Day +1 and +2 post-stem cell transfusion days
  * Cyclophosphamide on Days +3 and +4 post-transplant
  Interventions: Drug: Fludarabine; Radiation: Fractionated total body irradiation; Drug: Busulfan; Drug: Cyclophosphamide; Radiation: Single dose total body irradiation; Drug: Melphalan; Drug: Granulocyte-colony stimulating factor; Procedure: Stem cell transplant; Drug: Azacitidine

INTERVENTIONS:
Drug: Fludarabine
  Other Names: Fludara; 2-Fluoro-ara-A Monophosphate; 2-Fluoro-ara AMP; FAMP
Radiation: Fractionated total body irradiation
Drug: Busulfan
  Other Names: Myerlan; Busulphan
Drug: Cyclophosphamide
  Other Names: Cytoxan; CPM; CTX; CYT
Radiation: Single dose total body irradiation
Drug: Melphalan
  Other Names: Alkeran; Phenylalanine mustard
Drug: Granulocyte-colony stimulating factor
  Other Names: G-CSF; Plerixafor; Mozobil; Neupogen; Filgrastim
Procedure: Stem cell transplant
Drug: Azacitidine
  Other Names: Vidaza; Ladakamycin

SUMMARY:
Allogeneic hematopoietic cell transplantation (allo-HCT) is a potentially curative therapy for patients with hematologic malignancies including acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), and acute lymphoblastic leukemia (ALL); however, human leukocyte antigen (HLA)-matched donor availability continues to be a major hurdle. Historically, HLA haploidentical donor hematopoietic cell transplantation (haplo-HCT) was associated with high incidences of graft rejection and excessive non-relapse mortality (NRM), but recent advances utilizing post-transplant cyclophosphamide (PT-Cy) have revolutionized haplo-HCT and the outcomes are now comparable to allo-HCT using more traditional HLA matched related and unrelated donors. However, graft-versus-host disease (GvHD) continues to be a problem and is associated with significant morbidity and mortality in allo-HCT patients including those who receive haplo-HCT on PT-Cy platform. The aim of this early phase study is to investigate the safety and overall efficacy of azacitidine in reducing the incidence and severity of GvHD when added to PT-Cy based haplo-HCT platform for patients with AML, ALL, or advanced MDS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute leukemia (AML/ALL) or advanced MDS (INT-2 or high risk) in complete remission (CR/CRc/CRi) documented by bone marrow biopsy done within 30 days prior to the initiation of conditioning regimen.
* Available HLA-haploidentical donor that meets the following criteria:

  * Immediate family member (sibling, offspring, or parent)
  * At least 18 years of age
  * HLA-haploidentical donor/recipient match by class I serologic typing at the A&B locus.
  * In the treating physician's opinion, is in general good health, and medically able to tolerate leukapheresis required for harvesting HSC
  * No active hepatitis (B, C), HTLV, and HIV infections
  * Not pregnant
* Karnofsky performance status ≥ 70 %
* Adequate organ function as defined below:

  * Total bilirubin ≤ 2.5 mg/dl (unless the patient has a history of Gilbert's syndrome)
  * AST(SGOT) and ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ 2.0 x IULN OR estimated creatinine clearance ≥ 30 mL/min/1.73 m^2 by Cockcroft-Gault Formula
  * Oxygen saturation ≥ 90% on room air
  * LVEF ≥ 40%
  * FEV1 and FVC ≥ 50% predicted, corrected DLCO ≥ 40% predicted
* At least 18 years of age at the time of study registration
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* Recipients with donor sensitive antibodies (DSA), defined by 2000 or higher MFI against one or more class I or II antigens
* Known HIV or active Hepatitis B or C infection
* Underwent a previous related or unrelated allogeneic transplant
* Known hypersensitivity to one or more of the study agents
* Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of the conditioning regimen.
* Pregnant and/or breastfeeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or unstable cardiac arrhythmias.
* Presence of a readily available 6/6 matched sibling donor who is a candidate for donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Safety of azacitidine (Phase I only) as measured by frequency and grade of adverse events | Up to Day 35
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Maximum tolerated dose of azacitidine (Phase I only) | Estimated to be 3-4 months (completion of all Phase I patients through Day 35)
Grade II-IV acute GvHD rate of azacitidine (Phase II only) | Up to Day 100

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 48 months
  EFS is defined as the time from date of first dose of the preparative regimen until failure to engraft, treatment failure, disease progression/relapse, or death from any cause (whichever occurs first).
Overall survival (OS) | Up to 48 months
  OS is defined as the time from the date of Day 0 until death from any cause.
Disease-free survival (DFS) | Up to 48 months
Non-relapse mortality (NRM) | Up to Day 100
  NRM is defined as death that results from a transplant procedure-related complication (e.g. infection, organ failure, hemorrhage, GvHD) rather than from relapse of the underlying disease prior to Day +100 visit.
Time to neutrophil engraftment | Up to 12 months
  Time to neutrophil engraftment is measured by determining the first of 3 consecutive measurements of neutrophil count ≥ 500/ul following conditioning regimen-induced nadir.
Time to platelet engraftment | Up to 12 months
  Time to platelet engraftment is measured by determining the first of 3 consecutive measurements of platelet count ≥ 20,000/ul without platelet transfusion support for 7 days.
Rate of acute GvHD | Up to Day 100
  Incidence and severity of acute GvHD will be assessed based on the modified Glucksberg criteria and Seattle criteria. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Rate of chronic GvHD | Day 100 through Day 365
  Incidence and severity of chronic GvHD will be assessed based on the NIH consensus criteria and global severity scoring system. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu